CLINICAL TRIAL: NCT07210580
Title: Testing the Impact of Measurement-Based Care on Quality of Life and Disease Management Among Veterans With Inflammatory Bowel Disease: A Hybrid Effectiveness-Implementation Study
Brief Title: Testing the Impact of Measurement-Based Care on Quality of Life and Disease Management Among Veterans With Inflammatory Bowel Disease
Acronym: MBC-IBD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 24-026; 824-MR-48366 (Other Grant/Funding Number: Department of Veterans Affairs, HSR); 1845095 (Other: Central IRB)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease
Keywords: Measurement Based Care; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBC-IBD (Experimental): Measurement Based Care for Inflammatory Bowel Disease - Intervention group. Veteran participants who are randomized to 12-months of MBC-IBD will be enrolled for 12 months. They will each complete surveys at baseline, 6-months, and 12-months post-randomization. These assessments require completion of self-report questionnaires which will be completed by phone or electronically using VA REDCap. MBC in IBD will not replace but rather provide care continuity between clinic visits. Patients allocated to MBC in IBD will receive automated reminders to complete weekly questionnaires.
  Interventions: Behavioral: MBC-IBD Intervention
- E-TAU (Active Comparator): Enhanced Treatment as Usual (E-TAU). Participants assigned to E-TAU will receive standard of care, including monitoring and treatment as directed at the discretion of their gastroenterologist. Standard of care is based on current evidence-based professional guidelines, including routine inflammatory biomarker assessments (e.g., annual fecal calprotectin), therapy plans, scheduled and as-needed clinic visits, and scheduled and as-needed telephone calls. Participants will also receive educational videos and fact sheets on various IBD-specific topics.
  Interventions: Other: Enhanced Treatment as Usual (E-TAU)

INTERVENTIONS:
Behavioral: MBC-IBD Intervention — Measurement Based Care for Inflammatory Bowel Disease - Intervention group. Veteran participants who are randomized to 12-months of MBC-IBD will be enrolled for 12 months. They will each complete surveys at baseline, 6-months, and 12-months post-randomization. After baseline completion, participants will be asked to complete weekly surveys. These assessments require completion of self-report questionnaires (PROs) which will be completed by phone or electronically using VA REDCap. MBC in IBD will not replace but rather provide care continuity between clinic visits. Patients allocated to MBC in IBD will receive automated reminders to complete weekly questionnaires. Further, patients will receive quarterly reports of their PRO data trends.
  Arms: MBC-IBD
Other: Enhanced Treatment as Usual (E-TAU) — E-TAU will receive standard of care, including monitoring and treatment as directed at the discretion of their gastroenterologist. Participants will also receive educational videos and fact sheets on various IBD-specific topics.
  Arms: E-TAU

SUMMARY:
This research study is addressing issues related to Inflammatory bowel disease (IBD), which is a chronic autoimmune disorder that affects over 60,000 Veterans. With close monitoring and timely treatment adjustment, the investigators can stop the natural progression of IBD, improving health-related quality of life (HRQOL) and reducing flares and hospitalizations. However, it is difficult to closely monitor Veterans with IBD between clinic visits. There is a critical need for solutions that support close between visit monitoring of Veterans with IBD. The Measurement-Based Care (MBC) for IBD study will take a systematic approach to collect, share, and act on patient reported outcome (PRO) data that can be used to achieve close monitoring. MBC supports patients' in managing their condition and boosting their confidence in their ability to handle their symptoms and disease, and also supports care teams in early recognition of health issues. The investigators will work with both Veterans and their care teams to understand and assess this program so it can be a model for future initiatives.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic autoimmune disorder that affects over 60,000 Veterans and leads to highly symptomatic flares and complications. Close monitoring and timely treatment adjustment can stop the natural progression of IBD, improving health-related quality of life (HRQOL) and reducing flares and hospitalizations. However, it is difficult to closely monitor Veterans with IBD between clinic visits. There is a critical need for systematic solutions to support close between visit monitoring of Veterans with IBD without which they will continue to experience preventable impairment and disability. Measurement-based care (MBC) is a systematic approach to collect, share, and act on patient reported outcome (PRO) data that can be used to achieve close monitoring. MBC works by facilitating early recognition of clinical deterioration and timely clinician-driven treatment adjustment. MBC also increases patients' self-efficacy, their confidence in their ability to handle their symptoms and disease.

This project will use a Hybrid Type 1 effectiveness-implementation randomized trial design (n=250 Veterans with IBD) to test the effectiveness of MBC in IBD versus enhanced treatment as usual (E-TAU) on HRQOL and IBD-related events over 12-months and identify barriers and facilitators to MBC in IBD to inform its implementation in practice. The hypothesis is that at 12-month follow-up, Veterans randomized to MBC will have greater improvement in HRQOL and fewer IBD-related events (composite of flares, emergency department visits, hospitalization, surgery) than E-TAU. The primary objective is to test the effectiveness of MBC vs. E-TAU on key patient outcomes: IBD-specific patient reported HRQOL (primary outcome) and IBD-related events obtained via electronic health record data (secondary outcome). The secondary objective is to assess determinants of MBC in IBD implementation and acceptability with process evaluation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Veteran patients include:

* receiving IBD care at one of the four sites
* reporting an impaired IBD-specific HRQOL using the Short IBD Questionnaire (SIBDQ<60, as used by others)
* willingness and ability to participate in study procedures

Clinic staff criteria:

* relevant clinic staff (gastroenterologists, advanced practice providers, nurses) involved in MBC in IBD at the four study sites (Ann Arbor, Atlanta, Houston, Portland).

Exclusion Criteria:

Veteran Patient Exclusion criteria:

* Presence of an ostomy or ileal-pouch anal anastomosis
* Severe comorbid medical condition that can confound PRO scores and treatment priorities (e.g., cancer, transplant).
* Exclusions can be readily determined from chart review and a baseline patient assessment

Clinic staff exclusion criteria:

* Clinic staff without any experience with MBC in IBD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2028-12-29 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient-reported Health-related Quality of Life | Baseline compared to 12 month follow-up.
  Test the effectiveness of MBC vs. E-TAU on key patient outcomes, specifically looking at IBD-specific patient reported HRQOL (primary outcome).
  Assess IBD-specific HRQOL compared to E-TAU at 12-months follow-up. The investigators will first graphically explore the longitudinal data over time between the MBC and E-TAU groups. As the primary analytic model, the investigators will use an analysis of covariance (ANCOVA), fit using a linear regression model with SIBDQ score at 12 months as the dependent variable to estimate between-group differences in the primary endpoint. The model will include an indicator for treatment group (MBC vs. E-TAU) to estimate the 12-month treatment effect and adjust for baseline SIBDQ scores as a covariate and the stratification factors used for randomization (site, age, IBD type).

SECONDARY OUTCOMES:
IBD-related events | Baseline compared to 12 month follow-up.
  Review of IBD-related events obtained via electronic health record data: The investigators will first assess the total count of flares, emergency department visits, hospitalizations, and surgeries between baseline and 12 months and model cumulative composite outcomes at 12-months. If the total outcome counts are low (mostly 0's or 1's), the investigators will use a logistic regression model to model a dichotomized outcome. If the total counts have a range (e.g., 0 to 5 or more), the investigators will use a count data model such as Poisson or negative binomial regression model. The investigators will include intervention group (MBC vs. E-TAU) as the primary predictor, as well as study site, age, IBD type, and other covariates that show imbalances in baseline analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Cohen-Mekelburg, MD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (4):
- United States (4):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No